CLINICAL TRIAL: NCT03666663
Title: UCSF Sphenopalatine Ganglion Block Study- a Randomized Double Blind Placebo Controlled Trial to Compare Nasal Anesthetics for Migraine Prevention in Adults.
Brief Title: Sphenopalatine Ganglion Blocks RCT
Acronym: SPGblock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-25736_SPG_2018.09
Record Dates: First submitted 2018-09-08; First posted 2018-09-12 (Actual); Results first posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Lidocaine; Bupivacaine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lidocaine (Experimental): Participants will receive SPG blocks with lidocaine.
  Interventions: Drug: Lidocaine
- Bupivacaine (Experimental): Participants will receive SPG blocks with bupivacaine
  Interventions: Drug: Bupivacaine
- Ropivacaine (Experimental): Participants will receive SPG blocks with ropivacaine
  Interventions: Drug: Ropivacaine
- Placebo (saline) (Placebo Comparator): Participants will receive SPG blocks with placebo (saline)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — Nasal application using the Sphenocath device- cleared by FDA
  Arms: Lidocaine
Drug: Bupivacaine — Nasal application using the Sphenocath device- cleared by FDA
  Arms: Bupivacaine
Drug: Ropivacaine — Nasal application using the Sphenocath device- cleared by FDA
  Arms: Ropivacaine
Drug: Placebo — Placebo Saline using the Sphenocath device- cleared by FDA
  Other Names: Placebo Saline
  Arms: Placebo (saline)

SUMMARY:
RCT of Sphenopalatine Ganglion (SPG) Blocks using anesthetics vs. placebo for migraine.

DETAILED DESCRIPTION:
Chronic Migraine is a brain disorder with high prevalence. It is the 7th leading cause of disability worldwide according the WHO.

SPG block is a treatment for migraine that has been used for two decades. It can be done by needle injection of anesthetic to the region of the SPG. However, there are now multiple catheter devices that can be used to non-invasively administer anesthetic topically through the nasal cavity to the region of the SPG where the anesthetic is then absorbed through thin membranes covering the SPG.

Various anesthetic agents have been studied however currently, to our knowledge, there is no head to head comparison of the various anesthetics used. Studies of SPG blocks in the setting of chronic migraine are few as compared to the use of SPG as acute treatment for migraine.

With the use of an RCT, we aim to determine the overall efficacy of SPG blocks used at longer intervals than have been studied in the past as compared to placebo, as well as to examine the relative efficacy of the anesthetics used most commonly and studied for SPG blocks.

We will be using an FDA cleared device, the Sphenocath which was developed and registered with the FDA for this specific population and purpose. The study intervention is the standard practice in the UCSF Headache Center to perform SPG blocks for our patients with chronic migraine. The frequency we use in clinical practice and that we plan to study is less often than in previous studies of this intervention in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more at time of consent
2. Current patients in the UCSF Headache Center eligible to receive SPG blocks for migraine and would otherwise receive treatment clinically
3. Ability to provide consent for the research study

Exclusion Criteria

1. Pregnant or breast feeding within 4 weeks of enrollment
2. Inability to communicate with the study team
3. Patients who cannot read and understand English
4. Deemed unsuitable for enrollment in study by the investigator
5. Allergy to local anesthetics or saline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Riggins, MD, Principal Investigator — UCSF Headache Center
Locations (1):
- UCSF Headache Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goadsby PJ, Zagami AS, Lambert GA. Neural processing of craniovascular pain: a synthesis of the central structures involved in migraine. Headache. 1991 Jun;31(6):365-71. doi: 10.1111/j.1526-4610.1991.hed3106365.x. PMID 1889975
- [Background] Piagkou M, Demesticha T, Troupis T, Vlasis K, Skandalakis P, Makri A, Mazarakis A, Lappas D, Piagkos G, Johnson EO. The pterygopalatine ganglion and its role in various pain syndromes: from anatomy to clinical practice. Pain Pract. 2012 Jun;12(5):399-412. doi: 10.1111/j.1533-2500.2011.00507.x. Epub 2011 Sep 29. PMID 21956040
- [Background] Robbins MS, Robertson CE, Kaplan E, Ailani J, Charleston L 4th, Kuruvilla D, Blumenfeld A, Berliner R, Rosen NL, Duarte R, Vidwan J, Halker RB, Gill N, Ashkenazi A. The Sphenopalatine Ganglion: Anatomy, Pathophysiology, and Therapeutic Targeting in Headache. Headache. 2016 Feb;56(2):240-58. doi: 10.1111/head.12729. Epub 2015 Nov 30. PMID 26615983
- [Background] Mehta D, Leary MC, Yacoub HA, El-Hunjul M, Kincaid H, Koss V, Wachter K, Malizia D, Glassman B, Castaldo JE. The Effect of Regional Anesthetic Sphenopalatine Ganglion Block on Self-Reported Pain in Patients With Status Migrainosus. Headache. 2019 Jan;59(1):69-76. doi: 10.1111/head.13390. Epub 2018 Jul 25. PMID 30043973
- [Background] Binfalah M, Alghawi E, Shosha E, Alhilly A, Bakhiet M. Sphenopalatine Ganglion Block for the Treatment of Acute Migraine Headache. Pain Res Treat. 2018 May 7;2018:2516953. doi: 10.1155/2018/2516953. eCollection 2018. PMID 29862074
- [Background] Mojica J, Mo B, Ng A. Sphenopalatine Ganglion Block in the Management of Chronic Headaches. Curr Pain Headache Rep. 2017 Jun;21(6):27. doi: 10.1007/s11916-017-0626-8. PMID 28432602

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine | Bupivacaine | Ropivacaine | Placebo (Saline)
Started | 3 | 1 | 3 | 3
Completed | 3 | 1 | 1 | 1
Not Completed | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Bupivacaine | Ropivacaine | Placebo (Saline) | Total
Number analyzed (Participants) | 3 | 1 | 3 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 3 | 3 | 10
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 1 | 7
  Male | 1 | 0 | 0 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Headache Days From Baseline to Month 8 of Treatment
Description: Reduction in headache days from baseline to month 8 of treatment as self- reported by the patients (yes/no) and as per headache diary and retrospective charts review documentation
Time Frame: 8 months
Measure: Number; unit: participants
Arm/Group | Lidocaine | Bupivacaine | Ropivacaine | Placebo (Saline)
Number analyzed (Participants) | 3 | 1 | 3 | 3
participants | 3 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: follow up appointments and chart review
Arm/Group | Lidocaine | Bupivacaine | Ropivacaine | Placebo (Saline)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT03666663/Prot_SAP_000.pdf